CLINICAL TRIAL: NCT06384235
Title: An Open, Single-Arm, Phase II Clinical Study Evaluating the Efficacy and Safety of LTC004 Monotherapy in Patients With Metastatic Colorectal Cancer Who Have Failed Third-Line and Above Standard Treatment
Brief Title: Phase II Clinical Study of LTC004 in Patients With mCRC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Letolab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTC004-203
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Locally Advanced or Metastatic CRC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHASE 1 (Experimental): Enrollment of 10 consecutive evaluable CRC subjects with failure of existing standard therapy or lack of effective treatment Treated with LTC004 in Phase I
  Interventions: Drug: LTC004
- PHASE 2 (Experimental): If ≥2 subjects experience objective remission in PHASE 1, proceed to Phase II to enroll an additional 20 evaluable subjects to further evaluation of the safety and efficacy of LTC004
  Interventions: Drug: LTC004

INTERVENTIONS:
Drug: LTC004 — LTC004,45μg/kg,IV,Day 1,Q3W;

SUMMARY:
This is a phase II clinical study to evaluate the safety and antitumor activity of LTC004 in patients with locally advanced or metastatic CRC，Enrollment of 10 evaluable subjects in Phase I. If ≥2 subjects experience objective remission，proceed to Phase II to enroll an additional 20 evaluable subjects to further evaluation of the safety and efficacy of LTC004

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years.
2. Non-radical resectable metastatic colorectal cancer confirmed by histology or cytology (pathology report required).
3. Those who have progressed on, or are intolerant to, at least three lines of prior systemic antitumor therapy for metastatic colorectal cancer. Patients must have received fluorouracil, oxaliplatin, and irinotecan-based chemotherapy, as well as patients with mCRC who have received or are not candidates for prior anti-VEGF therapy, TKI agents, and anti-epidermal growth factor receptor therapy (RAS wild-type).
4. At least one measurable tumor lesion based on RECIST V1.1 criteria.
5. ECOG PS ≤1.
6. Expected survival ≥12 weeks.
7. Adequate organ function.
8. Patients, both females and males, of reproductive potential must agree to use adequate contraception during and for 6 months after the last infusion of LTC004.
9. Patients who have received any chemotherapy or anti-tumor monoclonal antibody drugs within 4 weeks prior to the first dose of study drug.small molecule targeted drugs within 2 weeks prior to the first dose of study drug; Chinese medicine therapy (Chinese medicine therapy with clear anti-tumor indications in the package insert within 4 weeks prior to the first dose of study drug.
10. Understands and provides written informed consent and willing to follow the requirements specified in protocol.

Exclusion Criteria:

1. History of severe hypersensitivity reactions to other mAbs.
2. Untreated, unstable or uncontrolled central nervous system (CNS) metastases with following exceptions:A. Clinically stable MRI scans and no progressive or uncontrolled neurologic symptoms or signs for at least 4 weeks prior to the first study treatment.
3. Tumor invasion of vital arteries resulting in high risk of bleeding, significant risk of perforation or already formed fistulae.
4. Patients with uncontrolled pleural effusion, pericardial effusion or abdominal effusion as judged by the investigator at screening.
5. Patients with untreated or clinically symptomatic spinal cord compression that has not been controlled.
6. Previous antitumor regimens include immunotherapy such as PD-1/L1 inhibitors, LAG3, TIGIT, IL-2, IL-15, CD3-like immunoagonists, and other cellular therapies.
7. ≥2 malignant tumors within 5 years prior to first dose of drug.
8. Moderate to severe dyspnea at rest, severe primary lung disease,current need for continuous oxygen therapy, or clinically active interstitial lung disease (ILD) or pneumonia due to advanced cancer or its complications; Grade ≥3 interstitial pneumonia during prior antineoplastic therapy.
9. Presence of severe infection within 4 weeks prior to first dose of medication.Presence of active infection requiring systemic antibiotic therapy with CTCAE grade ≥2 within 2 weeks prior to first dose.
10. History of serious cardiovascular disease.
11. Active bleeding disorders, including gastrointestinal bleeding, as evidenced by vomiting of blood, profuse hemoptysis, or black stools, have occurred in the 6 months prior to enrollment.
12. Active hepatitis B,hepatitis C infection,syphilis infection, active tuberculosis.
13. Patients with active, or previous autoimmune disease with potential for recurrence.
14. Immunodeficiency diseases or history of such diseases, including a positive serologic test for human immunodeficiency virus (HIV).
15. Arterial/venous thrombotic events within 6 months prior to the first dose of the drug.
16. Those who received radical radiation therapy within 4 weeks prior to the first dose and those who received palliative radiation within 14 days prior to the first dose.
17. Use of live or attenuated vaccines within 4 weeks prior to the first dose,or anticipated need for live or attenuated vaccines during the study period.
18. Major surgery (other than surgery for diagnostic purposes) within 4 weeks prior to the first dose, anticipation of major surgery (other than surgery for diagnostic purposes) during the study period, or diagnostic or low-invasive surgery within 7 days prior to the first dose (excluded for puncture biopsies).
19. Adverse effects of prior antitumor therapy have not recovered to CTCAE version 5.0 grade rating ≤1.
20. Patients who have received a previous allogeneic bone marrow/hematopoietic stem cell transplant or solid organ transplant.
21. Pregnant and lactating women.
22. Subjects who in the judgment of the investigator, have a history of other serious systemic disease or are unfit to participate in this trial for any other reason (the presence of psychiatric disorders in the patient that may affect compliance with the trial, alcohol, drug or substance abuse,etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2025-08-23 (Estimated); Study Completion 2025-08-23 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 12 months
  Antitumor efficacy of LTC004 treated CRC patients

SECONDARY OUTCOMES:
DOR | up to 12 months
  Duration of Response of LTC004 treated CRC patients
PFS | up to 12 months
  Progression-Free Survival of LTC004 treated sarcoma patients
OS | up to 12 months
  Overall Survival of LTC004 treated CRC patients

IPD SHARING:
Plan to Share IPD: No